CLINICAL TRIAL: NCT01335269
Title: An Open Label Phase I Dose Finding Study of BI 853520 Administered Orally in a Continuous Dosing Schedule in Patients With Various Advanced or Metastatic Non-hematologic Malignancies
Brief Title: A Study of BI 853520 in Patients With Various Types of Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1300.2; 2010-024609-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-07; First posted 2011-04-14 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Treatment arm (Experimental): BI 853520 once daily in a dose escalation schedule
  Interventions: Drug: BI 853520

INTERVENTIONS:
Drug: BI 853520 — BI 853520 once daily in a dose escalation schedule

SUMMARY:
The primary objective of this trial is to determine the safety and tolerability of BI 853520 monotherapy by defining the maximum tolerated dose (MTD) and recommending the dose for further trials in the development of this compound.

Secondary objectives are

* determination of the pharmacokinetic (PK) profile;
* exploratory pharmacodynamic analysis; and
* collection of preliminary data on anti-tumour efficacy.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria

1. Patients with a confirmed diagnosis of advanced, measurable or evaluable, nonresectable and/or metastatic non-hematologic malignancy, which has shown to be progressive in the last 6 months as demonstrated by serial imaging
2. Patients who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not amenable to established treatment options
3. Tumour tissue must be available for the determination of E-cadherin expression (archived tissue or fresh biopsy).
4. Recovery from reversible toxicities (alopecia excluded) of prior anti-cancer therapies (CTCAE grade < 2)
5. Age = 18 years
6. Life expectancy = 3 months
7. Written informed consent in accordance with International Conference on Harmonisation/Good Clinical Practice (ICH/GCP) and local legislation, including consent for PK samples, for using an archived tumour sample for determination of Ecadherin status, for reviewing previous tumour scans (and for providing skin biopsies, in patients in dose finding phase enrolled before protocol amendment 03)
8. Eastern Cooperative Oncology Group (ECOG), R01-0787) performance score 0-1

   Additional inclusion criteria in the expansion phase:
9. Patients must have measurable progressive disease within the last 6 months, according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria (version 1.1, R09-0262)
10. deleted
11. Patients must be willing to provide paired tumour biopsies for PD determination. Refer to section 5.6.3
12. Patients should fit into one of the categories described below:

I. Metastatic adenocarcinoma of the pancreas Patients should have preferably received at least one line of systemic treatment for metastatic disease and preferably not more than 2 prior regimens for metastatic disease.

II. Platinum-resistant ovarian carcinoma, defined as recurrence within 6 months after completion of prior platinum-based chemotherapy Patients should have received preferably no more than 5 previous lines of systemic treatment for metastatic disease.

III. Oesophageal carcinoma Patients with oesophageal carcinoma of adenocarcinoma- or squamous cell histology who have received preferably not more than 2 previous lines of systemic treatment for metastatic disease.

IV. Soft tissue sarcoma Patients should preferably have received no more than 2 previous lines of systemic treatment for metastatic disease.

Exclusion criteria:

* Serious concomitant non-oncological disease/illness
* Active/symptomatic brain metastases
* Second malignancy
* Pregnancy or breastfeeding
* Women or men who are sexually active and unwilling to use a medically acceptable method of contraception.
* Treatment with cytotoxic anti-cancer-therapies or investigational drugs within four weeks of the first treatment with the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determination of the MTD. It will be defined by the occurrence of dose-limiting toxicities (DLT) during the first treatment cycle of each patient in the dose finding phase | After the first 28 days of treatment

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) after first dose | up to 48 hours
AUCt,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose) | up to 48 hours
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) after the last dose in cycle 1 | up to 24 hours
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) after the last dose in cycle 1 | up to 24 hours
Disease control rate (CR or PR or SD per RECIST v1.1) ) | up to 39 months
Duration of disease control (measured from drug start date to the date of disease progression for patients who had CR or PR or SD during treatment) | up to 39 months
Objective response rate (CR or PR per RECIST v1.1) | up to 39 months
Tumour shrinkage (in millimetre) defined as change from baseline to the minimum post-baseline sum of diameters of target lesions. | up to 39 months
Pharmacodynamic assessment: phosphorylated and total PTK2 (FAK) modulation in tumour biopsies | baseline, day 22 and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Canada (2):
  - 1300.2.1002 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1300.2.1001 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- Netherlands (3):
  - 1300.2.31003 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1300.2.31001 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1300.2.31002 Boehringer Ingelheim Investigational Site, Utrecht

REFERENCES:
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000
- [Derived] de Jonge MJA, Steeghs N, Lolkema MP, Hotte SJ, Hirte HW, van der Biessen DAJ, Abdul Razak AR, De Vos FYFL, Verheijen RB, Schnell D, Pronk LC, Jansen M, Siu LL. Phase I Study of BI 853520, an Inhibitor of Focal Adhesion Kinase, in Patients with Advanced or Metastatic Nonhematologic Malignancies. Target Oncol. 2019 Feb;14(1):43-55. doi: 10.1007/s11523-018-00617-1. PMID 30756308
- [Derived] Verheijen RB, van der Biessen DAJ, Hotte SJ, Siu LL, Spreafico A, de Jonge MJA, Pronk LC, De Vos FYFL, Schnell D, Hirte HW, Steeghs N, Lolkema MP. Randomized, Open-Label, Crossover Studies Evaluating the Effect of Food and Liquid Formulation on the Pharmacokinetics of the Novel Focal Adhesion Kinase (FAK) Inhibitor BI 853520. Target Oncol. 2019 Feb;14(1):67-74. doi: 10.1007/s11523-018-00618-0. PMID 30742245